CLINICAL TRIAL: NCT06458842
Title: Postoperative Pain Protocol Limiting Narcotics for Laparoscopic Hand-assisted Donor Nephrectomy Patients: A Randomized Control Trial
Brief Title: Postoperative Pain Protocol Limiting Narcotics for Laparoscopic Hand-assisted Donor Nephrectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit desired number of patients in reasonable time frame
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, FRANK S. DARRAS MD, Principal investigator, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 495511
Record Dates: First submitted 2024-05-17; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Narcotic Use; Renal Transplant Donor of Left Kidney
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Patients in this group will receive ketamine, morphine PCA and caldolor for pain control
  Interventions: Drug: Ketamine
- placebo (Placebo Comparator): Patients in this group receive placebo, morphine PCA, and caldolor for pain control
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine
Other: Placebo
  Arms: placebo

SUMMARY:
Kidney donors represent healthy patients and their anticipated postoperative course should be uncomplicated and brief. This study looks to optimize the perioperative pain regimen of laparoscopic donor nephrectomy patients by minimizing or eliminating narcotics from the immediate post-operative period. Current postoperative standard of care after donor nephrectomy require narcotic analgesics. While narcotics are potent pain medications, they are often associated with complications including nausea, vomiting and dysfunction of the gastrointestinal tract causing prolonged complications.

The investigators seek to evaluate a peri-operative pain regimen limiting the usage of narcotics. This incorporates a perioperative analgesic course utilizing combination of an intravenous non-steroidal anti-inflammatory drug (NSAID), intravenous acetaminophen, and intravenous ketamine. All three have been demonstrated to be effective for the control of perioperative pain while decreasing narcotics use.

Prior to surgery, participants will be consented and randomly assigned to receive the standard of care perioperative pain management using intravenous narcotics as a patient-controlled analgesia (PCA) by itself plus placebo or along with the new protocol. The study will demonstrate it the new protocol will limit or eliminate the need for narcotics as a patient-controlled dose during the postoperative period.

Upon discharge from the hospital, patients will be followed in clinic and via home questionnaires annually for 5 years to evaluate satisfaction, renal function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* all individuals undergoing laparoscopic donor nephrectomies at Stony Brook Hospital

Exclusion Criteria:

* Patients excluded as a potential kidney donor or surgical candidate (renal failure, cancer, uncontrolled hypertension or diabetes, cognitively impaired adults, children, history of stroke, complicated coronary history or pregnant)
* Patients with a history of chronic pain or chronic pain medication use
* Patients who are undergoing open nephrectomies
* Allergy to NSAID or acetaminophen
* Hepatic disease or elevated transaminases
* Peptic Ulcer Disease
* Probenecid use
* History of traumatic brain injury
* Contraindications of Ketamine Use (recent head trauma, open eye injury or glaucoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | number of days immediately after the surgery
  length of stay after surgery

SECONDARY OUTCOMES:
post surgical complication rates | 30 day
postoperative renal function (serum creatinine) | up to 2 years after intervention
amount of narcotic pain medication use | starting immediately after the surgery, during the inpatient time period
postoperative nausea | number of patients reporting postoperative nausea during inpatient time period
return of bowel function (passage of flatus) | the number of days after surgery at which return of bowel function is achieved
date of postoperative ambulation | reported during inpatient time period

CONTACTS AND LOCATIONS:
Overall Officials: Frank Darras, MD, Principal Investigator — Stony Brook Medicine - Department of Urology

IPD SHARING:
Plan to Share IPD: No